CLINICAL TRIAL: NCT04254510
Title: The Effect of Myofascial Relaxation Technique on the Treatment of Primary Dysmenorrhea in Psoas Muscle
Brief Title: The Effect of Myofascial Release Technique on the Treatment of Primary Dysmenorrhea in Psoas Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, esra pehlivan, Principal investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRT_Dysmenorrhea
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-02

CONDITIONS: Woman; Primary Dysmenorrhoea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Myofascial relaxation technique
  Interventions: Other: Myofascial relaxation technique
- Control group (No Intervention)

INTERVENTIONS:
Other: Myofascial relaxation technique — * Before the intervention, the number of days of the last menstrual cycle of all participants, the number of painful days throughout the cycle, pain intensity values according to the Visual Analogue Scale will be recorded, and the scores will be recorded in the participants.
  * Technique of direct relaxation of fascia of both psoas muscles to the participants in the myofascial relaxation group since the end of the last cycle, 90-120 sec. It will be applied by the physiotherapist twice a week.
  Arms: Study Group

SUMMARY:
Dysmenorrhea is a series of pathological symptoms associated with menstruation that interfere with daily activities such as abdominal cramps and pain in the menstrual period. General symptoms such as nausea, vomiting, lumbago, diarrhea and headache are also common. Primary dysmenorrhea refers to menstrual pain that does not depend on the underlying pathology. The kidneys act on the fascia of the psoas muscle. If the psoas muscle does not shorten and grow sufficiently, the kidneys may not move for a certain period of time and may experience ptosis. This causes venous ponding and may cause varicocele in men and primary dysmenorrhea in women. Techniques to be applied directly to the fascia of the psoas muscle can reduce symptoms of dysmenorrhea in women. In the literature review, no studies investigating the effectiveness of a treatment applied directly and only on the psoas muscle on primary dysmenorrhea were not found. This study can set an example for future studies. In our study, myofascial relaxation technique will be applied in women with primary dysmenorrhoea and its effect on pain will be examined.

ELIGIBILITY:
Inclusion Criteria:

* The age range is 18-30,
* Intense pain compared to visual analog scale in the lower region of the abdomen during or just before the menstruation period (> 4),
* No pregnancy history,
* Not using drugs for dysmenorrhea symptoms

Exclusion Criteria:

* Not agreeing to participate in the study,
* Endometriosis, ovarian cyst, uterine fibroid, congenital malformation or pelvic inflammation,
* Having a diagnosis of secondary dysmenorrhea

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | 5 seconds
  Pain intensity will be questioned by scale.For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]) . To avoid clustering of scores around a preferred numeric value, numbers or verbal descriptors at intermediate points are not recommended

CONTACTS AND LOCATIONS:
Overall Officials: Tülay Ülkü Sevim, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- Esra Pehli̇van, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided